CLINICAL TRIAL: NCT06769282
Title: Cross-Cutting Trauma-Informed Peer Aggression and Dating Violence Prevention for Preteens Receiving Intensive Mental Health Services
Brief Title: Trauma-Informed Peer Aggression and Dating Violence Prevention for Preteens Receiving Intensive Mental Health Services
Acronym: SPARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K01CE003687 (NIH); K01CE003687 (NIH)
Record Dates: First submitted 2024-12-15; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Aggression Childhood; Teen Dating Violence
Keywords: Proactive and Reactive Aggression; Teen Dating Violence; Peer aggression; trauma; Adverse Childhood Experiences; partial hospitalization program
MeSH Terms: conditions — Wounds and Injuries | interventions — Methods; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (SPARE) plus Treatment as Usual (Experimental): Participants assigned to this arm will receive SPARE in the form of group therapy in addition to treatment as usual at a child partial program.
  Interventions: Behavioral: Experimental: Intervention (SPARE) plus Treatment as Usual
- Treatment As Usual (Active Comparator): Arm Description: Participants assigned to this arm will receive treatment as usual at a child partial program.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Experimental: Intervention (SPARE) plus Treatment as Usual — 5 components: (1) Social skills training, including selecting healthy friends and partners, (2) Problem solving with emphasis on positive outcomes of nonaggressive solutions, (3) Awareness of domineering behavior in self and conflict resolution skills, (4) emotion Regulation, and (5) psycho-education on ACEs and trauma. Each session will include 30 minutes of didactic instruction on the component with developmentally engaging activities to illustrate concepts and an individually tailored 15-minute narrative and mindfulness activity, which may address a traumatic memory depending on youth need and receptivity.
  Other Names: SPARE; Intervention (SPARE) plus Treatment as Usual
  Arms: Intervention (SPARE) plus Treatment as Usual
Behavioral: Treatment as Usual (TAU) — Treatment As Usual consists of individual, family, occupational, and art therapy, social skills and emotion regulation groups, and therapeutic milieu. All staff and clinicians are trained in the Incredible Years Parenting Program, which aims reduce behavioral problems, enhance children's social and emotional competence, and improve child-parent interactions. Children also receive individualized treatment tailored for their needs (e.g., sleep interventions). Behavioral health needs staff (BHS) facilitate children's skill acquisition and generalization, implement individualized behavior contingency programs, and assist caregivers with parenting strategies via daily check-ins
  Arms: Treatment As Usual

SUMMARY:
The goal of this clinical trial is to learn if this intervention (Social Skills, Problem Solving, emotion Regulation, and psycho-Education on Trauma: A Trauma-Informed Peer Aggression and Teen Dating Violence Prevention Program; SPARE) can treat peer aggression and prevent teen dating violence in preteens receiving intensive mental health services. The main questions it aims to answer are:

* Does receiving SPARE reduce proactive and reactive aggression at post-intervention and 3- and 9-month follow-ups?
* Does receiving SPARE reduce positive attitude about TDV, prevent TDV behaviors, and improve mental health outcomes at post-intervention and 3- and 9-month follow-ups?

Researchers will compare youth receiving SPARE to youth receiving treatment as usual to see if SPARE results in improved proactive and reactive aggression, TDV attitudes and behaviors, and mental health outcomes.

Participants will:

* Receive SPARE via group therapy incorporated into their daily programing at an intensive mental health program
* Complete study questionnaires at program intake and discharge as well as at 3-month and 9-month follow-up assessments

DETAILED DESCRIPTION:
SPARE will include 5 components: (1) Social skills training, including selecting healthy friends and partners, (2) Problem solving with emphasis on positive outcomes of nonaggressive solutions, (3) Awareness of domineering behavior and conflict resolution skills, (4) emotion Regulation, and (5) psycho-Education on ACEs and trauma. SPARE is group-based each of the 5 treatment components are designed to be delivered in two 45-minute sessions per week (see Table 3), for a total of 10 sessions. Each session will include 30 minutes of didactic instruction on the component with developmentally engaging activities to illustrate concepts and an individually tailored 15-minute narrative and mindfulness activity, which may address a traumatic memory depending on youth need and receptivity. SPARE will be delivered by the PI and will replace a social skills group twice a week at CP when it is implemented.

SPARE will be implemented in two sites of a child partial hospitalization program (A & B). Both sites CP serve youth 7-13 years old who (1) require services more intensive than outpatient care or (2) are transitioning from higher care (e.g., inpatient). Youth attend CP for 6 hours a day Monday through Friday. The modal length of stay for youth is 7 weeks. To minimize disruptions in CP care, SPARE will be implemented continuously at one site for 6 months (Active Phase) while TAU data is collected from the other site. After 6 months, conditions at each site will flip, resulting in approximately 5 cohorts of SPARE per site (n=88). Sites A and B will be randomly assigned using yoked randomization to Active Phase or TAU first. During Active Phase, all youth ≥11 years will receive SPARE two days per week (regardless of research eligibility).

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 11-13 years
* (2) enrolled in CP,
* (3) ability to write and speak in English
* (4) parent/guardian consent.

Exclusion Criteria:

* None

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Proactive and Reactive Aggression Questionnaire (PRA) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  6 items; 2 subscales to assess proactive and reactive aggression; preteen self-report and parent-report

SECONDARY OUTCOMES:
Acceptance of Couple Violence (ACV) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  11 items; 2 subscales that assess acceptance of male-to-female violence and female to male violence; preteen self-report
Conflict in Adolescent Dating and Relationship Inventory (CADRI) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  35 items; 5 subscales that assess physical abuse, relational abuse, sexual abuse, threatening behavior, verbal-emotional
Digital Relationship Behaviors (DRB) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  32 items; 4 subscales assessing victimization and perpetration of Threatening/Coercive Behavior and Monitoring Behavior
Children's Depression inventory (CDI-2) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  28 items for self-report; 17 items for parent report; Depression measure; preteen self-report; parent report
Screen for Child Anxiety Related Emotional Disorders (SCARED) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  41 items; 4 subscales that assess anxiety symptoms related to panic/somatic, generalized anxiety, separation, social, and school avoidance
Disruptive Behavior Disorders Scale | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  42 items; 4 subscales assessing symptoms of ADHD-Inattention, ADHD-Hyperactivity/Impulsivity, Conduct Disorder, and Oppositional Defiant Disorder; parent report
ABCD Substance Use Screener | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  10 items; 3 subscales assessing use of alcohol, tobacco, and marijuana; child report

OTHER OUTCOMES:
PROMIS Peer Relations-Short Form | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  8 items; 2 subscales assessing friendship quality and peer acceptance; preteen report; caregiver report
Problem-Solving Measure for Conflict (PSM-C). | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  6 items; Assesses problem solving skills, Child report
Conflict Resolution Style Inventory (CRSI) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  20 items; 5 subscales assessing styles of Competing, Avoiding, Accommodating, Compromising, and Collaborating; preteen report
Children's Emotion Management Scale (CEMS) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  33 items; 3 subscales assessing emotion regulation of anger, sadness, and worry; Child and parent report
Child and Adolescent Trauma Screen (CATS) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  40 items; 3 subscales assessing occurrence of potential traumatic event, trauma symptoms, and symptom impairment; child and parent report.
Domineering Awareness Questionnaire (AAQ) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  10 items; Assesses awareness of domineering behavior and aggression; child report
ACEs Knowledge Questionnaire (AKQ) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  10 items; Assesses knowledge of the impact on ACEs on relationships; child-report
Pubertal Development Scale (PDS) | Baseline, Termination of treatment at the child partial program (average of 7 weeks post-baseline), 3-month follow up, 9-month follow up
  5 items for boys; 6 items for girls; Assesses stage of pubertal development and onset of menarche (girls); child report

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Tampke, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data on preteens (i.e., 11- to 13-year-olds) who receive treatment at a child partial hospitalization program in the Northeast and their caregivers and who consent to participate in study research will be included.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The duration of preservation and sharing of the data will be a minimum of 10 years after the funding period. It will be stored in a HIPAA-compliant server at Rhode Island Hospital.
Access Criteria: Deidentified dataset will have free and public access. Data will be made available through the CDC repository.